CLINICAL TRIAL: NCT05467436
Title: Evaluation of Pharmacogenomics Testing to Precision Prescriptions in Periodontal Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, Ahmed El-Awady, Assistant Professor, Augusta University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 1490009
Record Dates: First submitted 2022-02-23; First posted 2022-07-20 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Oral Surgeries
Keywords: Pharmacogenomics; Precision prescriptions
MeSH Terms: interventions — Anesthetics, Local; Analgesics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): Subject will receive standard prescription for local anesthetics, IV sedation drugs and analgesics at the time of first surgery.
  Subject will receive individually tailored-prescription for local anesthetics, IV sedation drugs and analgesics, based upon pharmacogenomic assessment at the time of second surgery.
  Interventions: Drug: Local anesthetics, IV sedation drugs and analgesics.

INTERVENTIONS:
Drug: Local anesthetics, IV sedation drugs and analgesics. — Personalized prescription for local anesthetics, IV sedation drugs and analgesics, based on pharmacogenomic assesment, social, dietary and medication history

SUMMARY:
The different patients responses to medications vary from dose effectiveness to adverse drug reaction (ADRs). ADRs affect outpatient settings as it account for estimated 1 million emergency department visits and over 3.5 million physician office visits per year. This subsequently results in about 125,000 hospital admissions. Currently, genetic testing conclude recommendation of dose adjustment or drug stop. However, further step is needed toward individually tailored prescription plan. The purpose of this study is to determine if the efficacy of the genetic testing (Pharmacogenomics) combined with the dietary habits and medications history to design an individually tailored prescription plan. This individualized-prescriptions will be tested if to reduce adverse drug reaction and improve pain management in periodontal surgeries. Hence, the current study will recruit subjects planned for two periodontal surgeries and evaluate pain management during and after periodontal surgery as well as post-surgical complication with and without individually tailored prescription plan. In addition, a comparison will be performed on number of drugs added, stopped or had a dose adjustment.

DETAILED DESCRIPTION:
The objective of this study is to combine pharmacogenomics testing with social, dietary and medications history to formulate individualized-prescription plan and to test the effectiveness of this precession approach to reduce adverse drug reaction and improve pain management during and after periodontal surgeries.

The specific aims of the study are:

* Specific aim 1: To test the efficacy of combining pharmacogenomics, dietary habits as well as social and medical history data to tailor a personalized prescription for each periodontal patient.
* Specific aim 2: To determine the ability of personalized prescription to achieve more efficacious pain management during and after periodontal surgery. The study also aims to determine the effect of this approach in the adjustment of opioid dosages for these patients.
* Specific aim 3: To determine the effect of personalized prescription, using pharmacogenomics tool, on post-surgical complications related to medications.

Self-controlled case series (SCCS) design will be used for the study. After eligibility has been ascertained and consent has been obtained, subjects planned for 2 surgeries will be enrolled in the study. First surgery will be carried out with the standard prescription for medications. For the second surgery, medications will be prescribed based on individualized assessment and pharmacogenomics report for each subject. These medications will be prescribed based on a consult with the periodontal surgeon's and PhamD investigators of the study. Medications that will be assessed in the study are: local anesthetics, IV sedation drugs and analgesics.

ELIGIBILITY:
Inclusion Criteria:

* Subjects at least 18 years of age
* All potential subjects must sign an informed consent prior to study enrollment
* Subjects willing to receive a standard full-mouth periodontal examination
* Subjects planned for 2 or more periodontal surgeries.

Exclusion Criteria:

* Subjects with medical conditions that contraindicate periodontal surgeries. These medical condition include: recent myocardial infarction and cerebrovascular accident, recent valve prosthesis surgery, immunosuppression, uncontrolled bleeding disorders, active treatment of malignancy as well as intravenous bisphosphonate use.
* Subjects with back and neck injuries that will not allow them to be in supine position.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in subject-reported post-surgery pain levels | Average of pain ratings, recorded after each surgery in the first week after the surgery. Patient will receive 1 call every 2 days to report his/her pain scale. Patient will receive a total of 3 calls in the 1st week after surgery.
  Patient 's assessment of the pain on a scale of 0-10 in the first week after the surgery
Changes in post-surgery complications related to medications | Post-operative complication will be assessed 2-4 weeks after the surgery
  Post-operative complication will be classified for 6 grades.

SECONDARY OUTCOMES:
Changes in post-surgery sedation assessment | Evaluated by the surgeon at the same day of the surgery where sedation performed
  Evaluated using Riker Sedation-Agitation Scale

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed El-Awady, BDS, MS, PhD, Principal Investigator — Dental College of Georgia-Augusta University
Locations (1):
- Augusta University-Dental College of Georgia, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No